CLINICAL TRIAL: NCT07336693
Title: Changes in Bone Mineral Density and the Impact of Therapeutic Approaches in Postmenopausal Patients With Rheumatoid Arthritis
Brief Title: Bone Density Change in Postmenopausal Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Burak Ugur Cetin, MD, Istanbul University - Cerrahpasa
Other Study IDs: IstanbulUC-BCetin-03
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis (RA); Osteoporosis
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoporosis | interventions — Bone Density

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postmenopausal Patients with Rheumatoid Arthritis: Postmenopausal women with a confirmed diagnosis of RA were identified. Postmenopause was defined as ≥12 months of spontaneous amenorrhea or a prior bilateral oophorectomy; women receiving hormone replacement therapy who fulfilled these criteria were also considered postmenopausal.
  Interventions: Diagnostic Test: Bone Density Test

INTERVENTIONS:
Diagnostic Test: Bone Density Test — BMD values were obtained from DXA scans performed at the lumbar spine (L1-L4), femoral neck, and total femur. All DXA measurements were conducted at the Department of Nuclear Medicine using the same device, a Hologic QDR 4500SL (S/N 45624, Bedford, MA), to ensure methodological consistency. Reference values were based on the NHANES III.

SUMMARY:
Rheumatoid arthritis is associated with systemic inflammation-mediated bone loss, leading to an increased risk of osteoporosis and fractures, particularly in postmenopausal patients. Although disease-modifying antirheumatic drugs may help mitigate bone loss, comparative longitudinal data on different treatment strategies remain limited. This study aimed to evaluate changes in bone mineral density over time and assess the impact of conventional synthetic and biologic DMARDs, together with anti-osteoporotic therapy, on bone health.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with a confirmed diagnosis of rheumatoid arthritis

Exclusion Criteria:

* Concomitant inflammatory rheumatic diseases other than RA
* History of malignancy
* Uncontrolled or untreated endocrine or metabolic disorders affecting bone metabolism, such as primary hyperparathyroidism, Cushing's syndrome, severe renal failure, severe hepatic failure
* Incomplete medical records or missing data

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective study was conducted using patient data obtained from the electronic medical records of a university hospital over the past five years.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Bone Mineral Density | 1-2 years
  For each patient, the absolute values and changes in BMD between the two DXA time points for the lumbar spine, femoral neck, and total femur were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University - Cerrahpasa (IUC), Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Joffe I, Epstein S. Osteoporosis associated with rheumatoid arthritis: pathogenesis and management. Semin Arthritis Rheum. 1991 Feb;20(4):256-72. doi: 10.1016/0049-0172(91)90021-q. PMID 2042057
- [Background] Theander L, Willim M, Nilsson JA, Karlsson M, Akesson KE, Jacobsson LTH, Turesson C. Changes in bone mineral density over 10 years in patients with early rheumatoid arthritis. RMD Open. 2020 Feb;6(1):e001142. doi: 10.1136/rmdopen-2019-001142. PMID 32519976
- [Background] Kroot EJ, Nieuwenhuizen MG, de Waal Malefijt MC, van Riel PL, Pasker-de Jong PC, Laan RF. Change in bone mineral density in patients with rheumatoid arthritis during the first decade of the disease. Arthritis Rheum. 2001 Jun;44(6):1254-60. doi: 10.1002/1529-0131(200106)44:63.0.CO;2-G. PMID 11407683